CLINICAL TRIAL: NCT03154684
Title: Efficacy of the STARK Comprehensive Autonomy Health Care Package in Functional Recovery After a Hip Fracture: A Randomized Controlled Trial
Brief Title: Spitex-SpiTal-Autonomie-Reha-Kraft
Acronym: STARK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Recruitment
Sponsor: University of Zurich (Other)
Collaborators: Spitex Zürich, Switzerland (Unknown); City of Zurich, Switzerland (Unknown); University Hospital, Zürich (Other); University of Applied Sciences of Western Switzerland (Other); Ebnet Stiftung, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016-01820
Record Dates: First submitted 2017-05-04; First posted 2017-05-16 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Osteoporosis; Frailty; Hip Fractures
Keywords: Autonomy; Rehabilitation; Falls; Quality of life; Senior
MeSH Terms: conditions — Osteoporosis; Frailty; Hip Fractures | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STARK intervention (Active Comparator): New care concept for hip fracture patients
  Interventions: Other: STARK intervention
- Standard Care (Other): Swiss standard of care for hip fracture patients
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: STARK intervention — The STARK Intervention is a new care concept for hip fracture patients that enable hip fracture patient to return to their home directly after discharge from acute care. The STARK comprehensive autonomy health care package includes following services;
  * Multidisciplinary collaboration of geriatricians, nurses and Spitex (ambulant nursing service at home) starting already during acute care
  * Inspection of the environment at the patient's home
  * Care and autonomy support
  * Social life support
  * Secondary prevention strategies:
  * Home exercise program (3x/weeks)
  * Protein enriched food preparation (20g whey protein/day)
  * Support to take vitamin D supplementation (2000 IU/day)
  * Recommendation and support to eat calcium rich foods
  * Motivation to be physically active
  Arms: STARK intervention
Other: Standard of Care — Standard of Care involves inpatient rehabilitation or home-based or inpatient transitional nursing care
  Arms: Standard Care

SUMMARY:
The primary purpose of this study is to test if the STARK comprehensive autonomy health care package improves lower extremity function over time at 6 weeks, 3, 6 and 12 months after hip or pelvis fracture compared to the standard of care.

DETAILED DESCRIPTION:
Hip fractures are the most frequent and most severe fractures among seniors age 75 and older and they have severe consequences: After a hip fracture, 50% of older persons have permanent functional disabilities, 15-30% require long-term nursing home care, and 10-20% die within one year. Besides the personal burden, hip fractures account for substantial increasing health care expenses. Given the high prevalence, severity and cost of hip fractures, novel care concepts such as STARK are urgently needed to support functionality and autonomy of hip fracture patients - especially in for the first year after the fracture

The STARK Intervention is a new care concept for hip fracture patients, which was developed based on prior evidence from clinical trials performed at the Centre on Aging and Mobility at the University of Zurich and important interdisciplinary clinical expertise collected at the Geriatric Trauma Centre at the University Hospital Zurich, the Spitex Zürich, the Dept. of Geriatrics at the University Hospital Zurich, and the Federal Department of Health at the City of Zurich (Gesundheits- und Umweltsdepartement).

The aim of the STARK intervention is to enable hip fracture patient to return to their home directly after discharge from acute care by providing a high-quality care concept provided by an interdisciplinary team bridging acute Geriatric Care at the University Hospital and Spitex services (ambulant nursing service at home).

With this pilot study, the investigators want to test if the STARK comprehensive autonomy care package improves lower extremity function in the first year after a hip fracture compared to standard of care. Most important secondary outcomes are rate of falls, health care utilization, re-hospitalization and nursing home admission, as well as quality of life, cognitive function, bone mineral density and muscle mass in senior hip fracture patients.

This study will include 20 community-dwelling men and women aged 70+ who are hospitalized at the University Hospital Zurich or City Hospital Waid due to an acute hip or pelvis fracture and who are not capable to return home without help.

This is a randomized controlled pilot trial with two parallel groups including a control group receiving standard of care (inpatient rehabilitation or home-based or inpatient transitional nursing care) and an intervention group receiving the STARK comprehensive autonomy health care package. The STARK comprehensive autonomy health care package consists on one hand of the STARK-Spitex who will support the participants during the first three months at home and on the other hand of a secondary prevention program including home exercise (3x/week), protein enriched food preparation (20 g whey protein/day), motivation and recommendation for vitamin D supplementation(2000 IE/day), calcium intake and physical activity. The intervention starts already during acute care and involves a multidisciplinary team of geriatricians, nurses and Spitex who assess the care and utilities needs of the patient. Each study participant will undergo 5 clinical visits (at baseline, after 6 weeks, 3 months, 6 months, and 12 months). Between clinical visits, participants will be contacted by phone every month.

The STARK comprehensive autonomy health care package can contribute to a faster and sustainable recovery of autonomy after a hip fracture in seniors and might help to lower direct and indirect health care costs by reducing the number of re-hospitalization due to fall-associated injuries.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling prior to the hip fracture event
* Living alone or with a partner/family member
* Living in the city of Zurich
* age 70+
* Acute hip or pelvis fracture after minimal trauma (resulting from a fall occurring from a standard height and without the involvement of others or a vehicle)
* Living at home without or with minimal (i.e. no more than 1x/day) support from the Spitex (ambulant nursing service) before the hip fracture
* Participant is mentally competent (judicious) based on the treating physicians' opinion at the screening visit.
* Inpatient rehabilitation or inpatient transitional care at a nursing home or ambulatory standard of care
* The participant understands the study procedures and voluntarily agree to participate in the study and comply with all its procedures by giving written informed consent

Exclusion Criteria:

* Patients who are expected to return home without help (i.e. no more care than Spitex 1x/day or physiotherapy 2x/week needed) directly after acute care are excluded.
* Conservative treatment of acute hip fracture or surgical treatment that does not allow full weight bearing after surgery
* Currently under cancer treatment or has active cancer (except for non-melanoma skin cancer)
* Major visual or hearing impairment (visual and/or hearing aids are allowed) or other serious illness that would preclude participation
* 24-hour nursing care need as this cannot be offered within the STARK package
* Mobility impairment that precludes return to own apartment
* Planned nursing home admission after acute hospital stay
* Current participation in another clinical trial, or plans of such participation in the next 12 months (corresponding to the study duration)
* Inability to read and/or speak German to an extent necessary to understand instructions and participate in the study
* Unwilling to forego any additional vitamin D supplementation (bolus or regular intake).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Lower extremity function | 12 months
  Lower extremity function will be measured by the Short Physical Performance Battery (SPPB)

SECONDARY OUTCOMES:
Gait speed | 12 months
  Gait speed will be obtained from the SPPB.
Gait speed | 12 months
  Gait speed will be assessed by a 400 m walk test.
Grip strength | 12 months
  Hand grip strength will be measured using a Martin Vigorimeter.
Repeated sit-to-stand | 12 months
  Repeated chair stand test will be obtained from the SPPB.
Rate of falls | 12 months
  Rate of falls will be assessed by a monthly phone call.
Health care utilization | 12 months
  Health care utilization will be assessed using the health care utilization questionnaire.
Number of re-hospitalizations | 12 months
  All hospitalizations will be documented as part of the safety documentation(SAE).
Number of nursing home admissions | 12 months
  All nursing home admissions will be documented.
Adherence to preventive strategies | 3 months
  Adherence will be documented by the Spitex staff.
Adherence to preventive strategies | 12 months
  Adherence will be documented by an adherence questionnaire.
Quality of life | 12 months
  Quality of life will be assessed by the RAND SF-36 questionnaire.
Quality of life | 12 months
  Quality of life will be assessed by the EuroQol (EQ-5D-3L) questionnaire.
Cognitive function | 12 months
  Cognitive function will be assessed by the MoCA.
Cognitive function | 12 months
  Cognitive function will be assessed by the MMSE.
Appendicular muscle mass | 12 months
  Appendicular muscle mass will be assessed by dual energy X-ray absorptiometry.
Bone mineral density | 12 months
  Bone mineral density will be assessed by dual energy X-ray absorptiometry.
Activities of daily living | 12 months
  Activities of daily living will be assessed by questionnaire (PROMIS-HAQ)

OTHER OUTCOMES:
Interaction of family carer with hip-fracture patient and health professionals | 12 months
  The interaction will be assessed by semi-structured interviews with a family carer.

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff-Ferrari, Prof., Principal Investigator — Zentrum Alter und Mobilität
Locations (1):
- Dept. of Geriatrics and Aging Research, University of Zurich / Geriatric Clinic University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No